CLINICAL TRIAL: NCT05205538
Title: Does Biological Sex Influence the Cardiac Output Response to Sprint Interval Exercise Training in Humans?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Martin Gibala, Professor, McMaster University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 14279
Record Dates: First submitted 2021-12-23; First posted 2022-01-25 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Exercise
Keywords: Cardiac output
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Females (Experimental): Female participant group
  Interventions: Other: Sprint interval exercise training
- Males (Experimental): Male participant group
  Interventions: Other: Sprint interval exercise training

INTERVENTIONS:
Other: Sprint interval exercise training — A 10-minute sprint interval exercise training protocol that is performed three times per week for a total of 12 weeks.

SUMMARY:
Sprint interval exercise training refers to brief repeated bouts of vigorous effort that are separated by short periods of recovery. Cardiac output refers to the amount of blood that is pumped out of the heart each minute. Research has shown that sprint interval exercise training can increase peak cardiac output - or the highest cardiac output that is achieved during strenuous exercise - but this response may be influenced by biological sex. The primary goal of this study is to determine whether the peak cardiac output response to 12 weeks of sprint interval exercise training differs between males and females. Cardiac output will be estimated using a non-invasive technique that involves breathing in a mixture of standardized gases. This research will help to determine whether biological sex influences the response of the heart to brief vigorous cycle exercise training.

DETAILED DESCRIPTION:
The primary purpose of this study is to determine whether biological sex influences the peak cardiac output response to 12 weeks of sprint interval exercise training. Peak cardiac output will be determined non-invasively using an inert gas rebreathing technique. Each session of sprint interval exercise training will involve a 10-minute period of cycling on a stationary ergometer. The protocol will consist of a two-minute warm-up; three, 20-second 'all out' efforts that are separated by two minutes of recovery; and a three-minute cool down. Three sessions of training will be performed each week for a total of 12 weeks. Groups of male and female participants will be recruited and tested using best practice guidelines for sex-based comparisons of exercise responses. The study will advance knowledge regarding the potential for biological sex to influence the cardiovascular response to brief vigorous cycle exercise training.

ELIGIBILITY:
Inclusion Criteria:

* Being untrained based on a self-report of engaging in < 1 h of weekly moderate to vigorous physical activity based on the Canadian Society for Exercise Physiology Get Active Questionnaire.
* Having an estimated cardiorespiratory fitness in the lower 50% of adults in the specified age range based on the online fitness calculator available at: www.worldfitnesslevel.org.
* Females who are naturally cycling (i.e., not using any form of hormonal contraceptive) or are using a 2nd generation oral contraceptive.

Exclusion Criteria:

* Experiencing a condition that might preclude safe participation in physical activity and exercise, as determined by answering "Yes" to any question on Page 1 of the Canadian Society for Exercise Physiology Get Active Questionnaire.
* Females with a positive pregnancy test.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2022-01-25 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Peak cardiac output | Change from baseline after 12 weeks of sprint interval exercise training
  Peak cardiac output measured during exercise

SECONDARY OUTCOMES:
Peak oxygen uptake | Change from baseline after 12 weeks of sprint interval exercise training
  Peak oxygen uptake measured during exercise
Flow mediated dilation | Change from baseline after 4 and 12 weeks of sprint interval exercise training
  Brachial artery flow mediated dilation
Pulse wave velocity | Change from baseline after 4 and 12 weeks of sprint interval exercise training
  Central and peripheral pulse wave velocity

CONTACTS AND LOCATIONS:
Overall Officials: Martin Gibala, PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No